CLINICAL TRIAL: NCT00759655
Title: An Open-Label Study To Evaluate The Efficacy And Safety Of Xyntha In Children Less Than 6 Years Of Age In Usual Care Settings
Brief Title: Study Evaluating The Efficacy And Safety Of Xyntha In Children Less Than 6 Years Of Age
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-3315; B1831002 (Other: Pfizer); 3082B2-3315-WW
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2011-01-04 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Hemophilia A
Keywords: hemophilia A; Xyntha; ReFacto; moroctocog alfa; bleeding disorder
MeSH Terms: conditions — Hemophilia A; Hemostatic Disorders | interventions — recombinant factor VIII SQ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- open label (Other)
  Interventions: Biological: Moroctocog alfa

INTERVENTIONS:
Biological: Moroctocog alfa — Patients will receive Moroctocog alfa according to their investigator's prescription.

SUMMARY:
This study will be investigating the safety and efficacy of Xyntha (moroctocog alfa (AF-CC)) in male patients less than 6 years old. Annualized bleeding rates and physician / caregiver assessments of responses to treatment will be characterized. FVIII inhibitor levels will be assessed throughout the study.

DETAILED DESCRIPTION:
The study was terminated on 22 Sept 2009 due to competition with another Wyeth study for a similar patient population. The decision to terminate the trial was not based on any safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Male patients less than 6 years of age with moderately severe to severe hemophilia A (FVIII less than or equal to 2%).
* Treatment history of less than 50 exposure days to prior recombinant or plasma-derived FVIII replacement products.
* Not receiving treatment for HIV or hepatitis infection, or the patient is on a stable antiviral regimen at the time of enrollment in the study.

Exclusion Criteria:

* Presence of any bleeding disorder in addition to hemophilia A.
* Inhibitor titer of greater than or equal to 5 Bethesda Units (BU) at screening.
* Treated with immunomodulatory therapy during the screening period
* Treatment history of more than 5 exposure days (ED) to Xyntha.
* Known hypersensitivity to hamster protein.

Ages: 0 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-3315&StudyName=Study%20Evaluating%20The%20Efficacy%20And%20Safety%20Of%20Xyntha%20In%20Children%20Less%20Than%206%20Years%20Of%20Age

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to be conducted in major hemophilia centers in North America, Latin America, and Asia-Pacific regions. Seven (7) sites were initiated; however, recruitment occurred at only 1 site in United State of America (USA) between June 2009 to December 2009. The study was terminated by the Sponsor.
Groups:
- Xyntha: Participants received intravenous infusion (s) of Xyntha as per dosage and administration frequency as prescribed by the treating physician.
Period: Overall Study
Arm/Group | Xyntha
Started | 1
Completed | 0
Not Completed | 1
Not completed — Termination of the study by sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Xyntha
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: Month] | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Factor VIII (FVIII) Inhibitor Development
Description: Incidence of inhibitor development was defined as any result determined positive at a central laboratory (Bethesda inhibitor titer of >=0.6 BU/mL) using Nijmegen modification of the Bethesda assay.
Time Frame: Baseline to 24 months or early withdrawal.
Population: Intent-to-treat (ITT) population: Participants who had received at least 1 dose of Xyntha.
Measure: Number; unit: Percentage of participants
Arm/Group | Xyntha
Number analyzed (Participants) | 1
Percentage of participants | 0

2. Primary Outcome: Percentage of Participants With Less Than Expected Therapeutic Effects (LETE) in the On-Demand Setting
Description: LETE in the on-demand setting was based on the response to the treatment of a bleeding episode. LETE in the on-demand setting occurred if the participant recorded 2 successive "No Response" ratings (indicated there was no improvement at all between infusions or during the 24 hour interval following an infusion, or condition worsened) after 2 successive Xyntha infusions, respectively. The infusions was to be administered within 24 hours (=<24 hours) of each other for the treatment of the same bleeding event in the absence of confounding factor.
Time Frame: Baseline to 24 months or early withdrawal.
Population: The study was terminated, analysis was not conducted.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

3. Primary Outcome: Percentage of Participants With LETE in the Prophylaxis Setting
Description: The LETE in the prophylaxis setting was the occurrence of a bleed. LETE in the prophylaxis setting occurred if there was a spontaneous bleed within 48 hours (=<48 hours) after a regularly scheduled prophylactic dose of Xyntha (which was not used to treat a bleed) in the absence of confounding factors.
Time Frame: Baseline to 24 months or early withdrawal.
Population: The study was terminated, analysis was not conducted.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

4. Primary Outcome: Percentage of Participants With Low Recovery LETE
Description: The LETE could be considered lower than expected recovery of FVIII in the opinion of the investigator following infusion of Xyntha in the absence of confounding factors.
Time Frame: Baseline to 24 months or early withdrawal.
Population: The study was terminated, analysis was not conducted.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

5. Secondary Outcome: Mean Annualized Bleed Rate (ABR)
Description: An annualized bleeding rate (ABR) for each participant was calculated as the number of bleeds requiring administration of FVIII replacement product (taken from the electronic Infusion Log Diary), divided by his total therapy duration (in days), and then multiplied by 365.25.
Time Frame: Baseline to 24 months or early withdrawal.
Population: The study was terminated, analysis was not conducted.
Units Other Than Participants: Bleeds
Arm/Group | Xyntha
Number analyzed (Participants) | 0
Number analyzed (Bleeds) | 0

6. Secondary Outcome: Number of Xyntha Infusions Needed to Treat Each New Bleed
Description: The data from the electronic Infusion Log Diary plus the Test Article case report form (CRF) was used to determine the number of infusions administered to treat a bleed. This was calculated by adding the initial 'for a new bleed' (on demand) infusion to any subsequent (on demand) infusions for the (same) 'previously treated bleed'. An on-demand infusion for a 'previously treated bleed' was counted toward the bleed with the most recent start time prior to that infusion.
Time Frame: Baseline to 24 months or early withdrawal.
Population: The study was terminated, analysis was not conducted.
Units Other Than Participants: Number of Infusions
Arm/Group | Xyntha
Number analyzed (Participants) | 0
Number analyzed (Number of Infusions) | 0

7. Secondary Outcome: Response to First On-demand Xyntha Treatment for All New Bleeds as Assessed by the Caregiver
Description: A 4-point response scale to be completed is as defined as follows: (Excellent: definite pain relief/improvement in signs of bleeding starting within 8 hrs after an infusion, with no additional infusion; Good: definite pain relief/improvement in signs of bleeding starting within 8 hrs or following the infusion; Moderate: probable/slight improvement starting after 8 hours following the infusion; No Response: no improvement at all between infusions).
Time Frame: Baseline to 24 months or early withdrawal
Population: The study was terminated, analysis was not conducted.
Arm/Group | Xyntha
Number analyzed (Participants) | 0

8. Secondary Outcome: Mean Number of Breakthrough (Spontaneous/Non-traumatic) Bleeds
Description: The number of breakthrough (spontaneous/non-traumatic) bleeds within 48 hours following a prophylaxis dose of Xyntha was summarized. The data from the electronic Infusion Log Diary plus the Test Article CRF was used to determine the number of infusions administered to treat a new bleed, counting only those infusions administered =<48 hours after an infusion marked as 'prophylaxis' (which had no associated bleed).
Time Frame: Baseline to 24 months or early withdrawal.
Population: The study was terminated, analysis was not conducted.
Units Other Than Participants: Bleeds
Arm/Group | Xyntha
Number analyzed (Participants) | 0
Number analyzed (Bleeds) | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the signing of the informed consent form to minimum 15 days after the last administered dose of Xyntha.
Description: Safety population = subjects who received at least 1 dose of Xyntha. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Xyntha
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyntha (N=1)
Anal fistula (Gastrointestinal disorders) | 1 (2)
Anal abscess (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xyntha (N=1)
Infusion site extravasation (General disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2)
Haematoma (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.